CLINICAL TRIAL: NCT01813708
Title: The Effectiveness of an Intensive Life-Style Intervention Compared to an Collaborative Educational Intervention On Metabolic Control, and Its Impact on Weight, Physical Activity, Quality of Life, Self-Efficacy in Type 2 Diabetes Patients
Brief Title: Intensive Life-Style Intervention in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mireya Gamiochipi Cano, MSc, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-716-0107
Record Dates: First submitted 2012-06-18; First posted 2013-03-19 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Intensive Life-Style; Collaborative Education; Clinical Trial; Metabolic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Life-Style Counseling (Experimental): 16 weekly sessions conducted by certified nutritionists certified in behavioural modification, and self-care techniques, including self-monitoring, healthy nutrition, physical activity, problem solving, relapse prevention, self-reinforcement, long-term motivation, and stress management
  Interventions: Behavioral: Intensive Life-Style
- Collaborative Educational (Active Comparator): 16 weekly sessions conducted by certified diabetes educators including: diabetes knowledge, nutrition, exercise, goal establishment in diabetes, problem solving, relapse prevention, self-monitoring, family and sexuality in diabetes, emotional management in diabetes, and stress management. Patients established their own goals
  Interventions: Behavioral: Collaborative Education

INTERVENTIONS:
Behavioral: Intensive Life-Style — 16 weekly sessions conducted by certified nutritionists certified in behavioural modification, and self-care techniques, including self-monitoring, healthy nutrition, physical activity, problem solving, relapse prevention, self-reinforcement, long-term motivation, and stress management
  Arms: Intensive Life-Style Counseling
Behavioral: Collaborative Education — 16 weekly sessions conducted by certified diabetes educators including: diabetes knowledge, nutrition, exercise, goal establishment in diabetes, problem solving, relapse prevention, self-monitoring, family and sexuality in diabetes, emotional management in diabetes, and stress management. Patients established their own goals
  Arms: Collaborative Educational

SUMMARY:
200 type 2 diabetes patients will be randomly submitted to an intensive life-style or a collaborative educational programmes by means of random numbers list. The intervention will be conducted by certified nutritionists or certified diabetes educators, previously trained in behavioural modification and in self-care techniques. The intervention will last 16 weekly sessions and A1c, LDL cholesterol, blood pressure will be measured as main variables. Furthermore, body weight and abdominal girth, other lipids (HDL cholesterol, triglycerides),and physical activity, quality of life, psychological well-being and self-efficacy will be measured with specific questionnaires for up to 6 months.

DETAILED DESCRIPTION:
Two interventions will be compared for metabolic control (A1c, LDL Cholesterol, and blood pressure). Additional measures will include: body weight abdominal girdle, other lipids (HDL cholesterol, triglycerides);and physical activity, quality of life, psychological well-being and self-efficacy will be measured with specific questionnaires.

Inclusion criteria are: Type 2 diabetes (ADA criteria) diagnosed during the last 3 years, without chronic complications, negative urine ketone tests, current in their dues to IMSS, A1c > 7%, and BMI > 25. No age limits.

Exclusion criteria: Psychosis or personality disorders, other illnesses thought to be fatal in 6 months or less (e.g. AIDS, liver Cirrhosis, etc), unable to read and write, and currently taking other drugs that impair blood glucose metabolism, such as glucocorticoids. Patients unable to perform physical activity because of other neurological, orthopedic or rheumatological conditions, patients on drug treatment for depression or obesity. Patients with alcohol or other drug dependencies, and being a relative of a patient already included in the study.

Patients will be randomly assigned to either intervention and will not be told to which intervention he/she was assigned.

The Intensive intervention is structured in 16 sessions to be held every week for groups of up to 15 patients in family medicine clinics in Mexico City. This includes healthy nutrition and physical activity plus behavioural modification techniques; the treatment goals will be instituted by the case manager (lowering body weight by 5% 10%, and increasing physical activity to 150 minutes/week).

The Educational Collaborative group will attend 16 weekly sessions where nutritional and physical activity will also be discussed, along with knowledge about diabetes and its treatment. Behavioural modification techniques are included in the curricula but the treatment goals will be selected by the patients themselves.

Blood samples will be drawn from an antecubital vein before the program starts and every 3 months thereafter. Measurements will include: A1c, glucose, total cholesterol, LDL, HDL cholesterol and triglycerides. Furthermore, body weight and abdominal girdle will be measured by a trained nurse observer who does not know the patient's group allocation. Questionnaires for physical activity, quality of life, psychological well-being and self-efficacy will be answered by patients every 3 months.

The statistical analysis will be conducted as an intention-to-treat analysis, and will include comparison of proportions of patients attaining treatment goals, adjusted by age, sex, BMI, and base-line values with logistic regression; continuous variables will be analyzed with Analysis of Covariance.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (ADA criteria) diagnosed during the last 3 years. Without chronic complications, negative urine ketone tests, current in their dues to IMSS, A1c > 7%, and BMI > 25. No age limits.

Exclusion Criteria:

* Psychosis or personality disorders, other illnesses thought to be fatal in 6 months or less (e.g. AIDS, liver Cirrhosis, etc), unable to read and write, and currently taking other drugs that impair blood glucose metabolism, such as glucocorticoids.
* Patients unable to perform physical activity because of other neurological, orthopedic or rheumatological conditions, patients on drug treatment for depression or obesity.
* Patients with alcohol or other drug dependencies, and being a relative of a patient already included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
disease control | 6 months
  Proportion of patients attaining pre-specified goals:
  A1c < 7%, LDL cholesterol < 100 mg/dl, blood pressure < 130/80 mmHg.

SECONDARY OUTCOMES:
Body Weight | 6 months
  Body Weight, reduction in abdominal girdle,HDL, Triglycerides
Quality of Life | 6 months
  Quality of life as assessed by the Jacobson Diabetes Quality of Life Measure
Well-Being | 6 months
  Well-being by the 22 item Bradleys Well-Being Questionnaire
Self-Efficacy | 6 months
  Self Efficacy with the Attitudes in Diabetes Questionnaire of Anderson, Funnel, Fitzgerald and Marrero

CONTACTS AND LOCATIONS:
Overall Officials: Niels H Wacher, MD, MSc, Study Chair — Instituto Mexicano del Seguro Social; Mireya Gamiochipi, MSC, Principal Investigator — Coordinación de Investigación en Salud, Mexico
Locations (1):
- Unidad de Investigación en Epidemiología Clínica, UMAE Hospital de Especialidades, Centro Médico Siglo XXI, IMSS, Mexico City, Mexico City, Mexico